CLINICAL TRIAL: NCT03646773
Title: Microvascular Effects of Intravenous Esmolol in Patients With Normal Cardiac Function Undergoing Postoperative Atrial Fibrillation: a Prospective Pilot Study in Cardiothoracic Surgery
Brief Title: Microvascular Effects of Intravenous Esmolol During Postoperative Atrial Fibrillation
Acronym: FANI
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0743_1
Record Dates: First submitted 2018-08-14; First posted 2018-08-24 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Postoperative Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Postoperative atrial fibrillation (POAF) is commonplace after cardiothoracic surgery. A rate control strategy by using short-acting beta blockers is recommended as a first-line therapy in patients without hemodynamic instability. Microcirculatory effects of POAF and esmolol have not been yet investigated. The investigators made the hypothesis that POAF without hemodynamic instability would induce microvascular dysfunction which could be reversed by intravenous esmolol.

ELIGIBILITY:
Inclusion Criteria:

* conventional cardiac surgery
* thoracic surgery

Exclusion Criteria:

* Postoperative atrial fibrillation leading to hemodynamic instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled for conventional cardiac or thoracic surgery who experienced in-hospital postoperative atrial fibrillation within the first seven postoperative days
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
effects of POAF without hemodynamic instability on near infrared spectroscopy (NIRS) parameters in combination with a vascular occlusion test | Day 7
  NIRS parameters were restoration speed and desaturation speed. Desaturation speed and resaturation speed of the study were assessed during POAF without esmolol and after a stabilization period of 45 min between each dose of esmolol. An automated pneumatic cuff inflator was positioned at the upper extremity of the ipsilateral upper limb. After completion of a baseline set of measurements for each patient, a rapid arterial occlusion of the upper limb was provoked by inflation of the pneumatic cuff at 50 mmHg above the systolic arterial pressure, up to the StO2 value decreases to 40% or for a maximal period of 10 minutes. The arterial cuff was then rapidly deflated to initiate reperfusion.